CLINICAL TRIAL: NCT04000360
Title: Pragmatic Cyclical Lower Extremity Exercise Trial for Parkinson's Disease
Acronym: CYCLE-II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH); University of Utah (Other)
Responsible Party: Principal Investigator, Jay Alberts, Principal Investigator, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2R01NS073717-06A1 (NIH); 2R01NS073717-06A1 (NIH)
Record Dates: First submitted 2019-06-25; First posted 2019-06-27 (Actual); Results first posted 2025-06-18 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Parkinson Disease
Keywords: Exercise
MeSH Terms: conditions — Parkinson Disease; Motor Activity

STUDY DESIGN:
Intervention Model Description: 252 mild to moderate PD patients will be randomized into a home cycling high-intensity aerobic exercise (AE) group or a Usual and Customary Care (UCC) group, asked to continue normal activity level and not initiate a formal cycling program during study participation.
Who Masked: Outcomes Assessor
Masking Description: The Movement Disorders Society Unified Parkinson's Disease Rating Scale (MDS-UPDRS III) will be conducted by a consistent rater, blinded as to participant randomization group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-Intensity Exercise Group (Experimental): Mild to moderate Parkinson's disease patients: The exercise group will be asked to cycle 3x/week for 12 months on a Peloton bicycle which will be delivered to their home.
  Interventions: Other: High-Intensity Aerobic Exercise (AE)
- Usual and Customary Care Group (Other): Mild to moderate Parkinson's disease patients, receiving no exercise intervention through the research but monitored with a parallel attention control. They will continue to receive usual and customary care for their Parkinson's disease during the 12 month period.
  Interventions: Other: Usual and Customary Care (UCC)

INTERVENTIONS:
Other: High-Intensity Aerobic Exercise (AE) — The home-based exercise group will have a Peloton indoor cycle, heart rate monitor strap, and Garmin activity monitor to track daily activity levels delivered to the home. Participants will be asked to cycle 3x/week for 12 months on this bike with heart rate monitor at aerobic intensity 60-80% of heart rate reserve and target cadence 80-90 revolutions per minute. Study team members will telephone all participants biweekly for similar contact times between treatment groups. During these calls, a study team member reviews fall diary information, inquires about possible adverse events, and reviews participants' activity monitor wear times on the Garmin Connect website (https://connect.garmin.com). For those in the AE group, exercise recommendations, e.g., increase duration, cadence or heart rate, are given based on review of exercise session data on the Peloton portal (onepeloton.com). Compliance barriers or technical challenges with the activity monitor or exercise cycle are addressed.
  Arms: High-Intensity Exercise Group
Other: Usual and Customary Care (UCC) — Participants in this group will continue to receive their usual care. They will also receive activity monitors to monitor their daily activity levels, and telephone monitoring throughout the study. Study team members telephone all participants every 2 weeks for similar amounts of contact time between treatment groups. During the calls, a study team member of the reviews fall diary information, inquires about possible adverse events, and reviews participants' activity monitor wear times via the Garmin Connect website (https://connect.garmin.com).
  Arms: Usual and Customary Care Group

SUMMARY:
Identification of an effective disease-modifying intervention (e.g. pharmaceutical, surgical or behavioral) is an unmet need in Parkinson's disease (PD). Increasing evidence indicates high intensity aerobic exercise is a candidate to alter PD progression. The primary aim of this study is to examine the disease-altering capabilities of a long-term, high-intensity aerobic exercise intervention. A multi-site pragmatic randomized controlled trial design has been selected. Individuals with PD will be randomized into 1) a home-based aerobic exercise program, or 2) a usual and customary care (UCC). Subjects in the home exercise group will receive an indoor stationary bicycle delivered to their home for a 12 month exercise period. Individuals in the UCC group will continue their current level of physical activity. Motor and non-motor assessments will be conducted at the main campus of the Cleveland Clinic or the University of Utah at enrollment, 6 months, and 12 months. Each assessment will last approximately one hour.

DETAILED DESCRIPTION:
Overview of Experimental Design: The study is a randomized controlled clinical trial designed to examine the disease-altering capabilities of a 12 month aerobic exercise program for individuals with PD. A total of 252 individuals with PD will be randomized into 1) a home-based aerobic exercise program, or 2) a usual and customary care (UCC). Subjects in the home exercise group will receive a commercially available Peloton indoor stationary bicycle delivered to their home for a 12 month exercise period. Individuals in the UCC group will continue their current level of physical activity. Both groups will undergo a series of motor and non-motor assessments at enrollment, 6 months, and 12 months to measure disease progression of the 12 month period. Additionally, data will be used to develop a prognostic model to predict 12-month change in Movement Disorder Society - Unified Parkinson's Disease Rating Scale III (MDS-UPDRS III) for patients participating in a home-based high-intensity aerobic exercise program.

ELIGIBILITY:
Inclusion Criteria:

* Adult with a diagnosis of idiopathic PD by a physician or physician extender
* Hoehn and Yahr stage I-III
* Demonstrate the ability to safely mount and dismount the Peloton stationary cycle
* In-home wireless network (WiFi; required for Peloton system exercise data transmission)

Exclusion Criteria:

* Participation in pharmaceutical or behavioral disease modifying PD-related clinical trial or study
* Diagnosis of dementia or any neurocognitive impairment that compromises one's ability to provide informed consent
* Implanted deep brain stimulation electrodes
* If the American College of Sports Medicine (ACSM) screen recommends medical clearance, the subject must obtain medical clearance by their health care provider prior to participation.
* Any musculoskeletal issue that would limit one's ability to engage in exercise
* Neurological disease other than Parkinson's disease (i.e. multiple sclerosis, stroke)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 256 (Actual)
Dates: Start 2019-11-13 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jay L Alberts, PhD, Principal Investigator — The Cleveland Clinic
Locations (2):
- United States (2):
  - Cleveland Clinic, Cleveland, Ohio
  - University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rudick RA, Miller D, Bethoux F, Rao SM, Lee JC, Stough D, Reece C, Schindler D, Mamone B, Alberts J. The Multiple Sclerosis Performance Test (MSPT): an iPad-based disability assessment tool. J Vis Exp. 2014 Jun 30;(88):e51318. doi: 10.3791/51318. PMID 25046650
- [Background] Rhodes JK, Schindler D, Rao SM, Venegas F, Bruzik ET, Gabel W, Williams JR, Phillips GA, Mullen CC, Freiburger JL, Mourany L, Reece C, Miller DM, Bethoux F, Bermel RA, Krupp LB, Mowry EM, Alberts J, Rudick RA. Multiple Sclerosis Performance Test: Technical Development and Usability. Adv Ther. 2019 Jul;36(7):1741-1755. doi: 10.1007/s12325-019-00958-x. Epub 2019 May 3. PMID 31054035
- [Background] Rosenfeldt AB, Penko AL, Jansen AE, Lopez-Lennon C, Zimmerman E, Imrey PB, Singh TK, Dibble LE, Alberts JL. Refining Maximal Heart Rate Estimation to Enhance Exercise Recommendations for Persons With Parkinson Disease. Arch Phys Med Rehabil. 2025 Nov;106(11):1680-1684. doi: 10.1016/j.apmr.2025.03.046. Epub 2025 Apr 5. PMID 40194736
- [Background] Alberts JL, Rosenfeldt AB, Lopez-Lennon C, Suttman E, Jansen AE, Imrey PB, Dibble LE. Effectiveness of a Long-Term, Home-Based Aerobic Exercise Intervention on Slowing the Progression of Parkinson Disease: Design of the Cyclical Lower Extremity Exercise for Parkinson Disease II (CYCLE-II) Study. Phys Ther. 2021 Nov 1;101(11):pzab191. doi: 10.1093/ptj/pzab191. PMID 34363478
- [Background] Rao SM, Losinski G, Mourany L, Schindler D, Mamone B, Reece C, Kemeny D, Narayanan S, Miller DM, Bethoux F, Bermel RA, Rudick R, Alberts J. Processing speed test: Validation of a self-administered, iPad(R)-based tool for screening cognitive dysfunction in a clinic setting. Mult Scler. 2017 Dec;23(14):1929-1937. doi: 10.1177/1352458516688955. Epub 2017 Jan 12. PMID 28080262
- [Background] Alberts JL, Rosenfeldt AB. The Universal Prescription for Parkinson's Disease: Exercise. J Parkinsons Dis. 2020;10(s1):S21-S27. doi: 10.3233/JPD-202100. PMID 32925109
- [Result] Jansen AE, Rosenfeldt AB, Lopez-Lennon C, Fernandez H, Zimmerman E, Imrey PB, Dibble LE, Alberts JL. Characterizing Hand Function in Parkinson's Disease Patients with a Self-Administered Electronic Manual Dexterity Test. Mov Disord Clin Pract. 2025 Mar;12(3):333-339. doi: 10.1002/mdc3.14286. Epub 2024 Nov 27. PMID 39604309
- [Result] Rosenfeldt AB, Jansen AE, Lopez-Lennon C, Zimmerman E, Imrey PB, Dibble LE, Alberts JL. Physical Activity Declines over a 12-Month Period in Parkinson's Disease: Considerations for Longitudinal Activity Monitoring. Med Sci Sports Exerc. 2025 Apr 1;57(4):738-745. doi: 10.1249/MSS.0000000000003615. Epub 2024 Nov 26. PMID 39589012
- [Result] Anis S, Zimmerman E, Jansen AE, Kaya RD, Fernandez HH, Lopez-Lennon C, Dibble LE, Rosenfeldt AB, Alberts JL. Cognitive measures predict falls in Parkinson's disease: Insights from the CYCLE-II cohort. Parkinsonism Relat Disord. 2025 Apr;133:107328. doi: 10.1016/j.parkreldis.2025.107328. Epub 2025 Feb 11. PMID 39956037
- [Result] Rosenfeldt AB, Lopez-Lennon C, Suttman E, Jansen AE, Owen K, Dibble LE, Alberts JL. Use of a Home-Based, Commercial Exercise Platform to Remotely Monitor Aerobic Exercise Adherence and Intensity in People With Parkinson Disease. Phys Ther. 2024 Feb 1;104(2):pzad174. doi: 10.1093/ptj/pzad174. PMID 38206881
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2024 Apr 8;4(4):CD013856. doi: 10.1002/14651858.CD013856.pub3. PMID 38588457
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2023 Jan 5;1(1):CD013856. doi: 10.1002/14651858.CD013856.pub2. PMID 36602886

RESULTS

PARTICIPANT FLOW:
Groups:
- Aerobic Exercise Group: Aerobic Exercise on a Stationary Bike
- Usual and Customary Care Group: Continue regular activity. No aerobic exercise intervention.
Period: Overall Study
Arm/Group | Aerobic Exercise Group | Usual and Customary Care Group
Started | 129 | 127
Completed | 123 | 123
Not Completed | 6 | 4

BASELINE CHARACTERISTICS:
Population: Mild to moderate Parkinson's disease patients
Groups:
- High-Intensity Aerobic Exercise Group: Mild to moderate Parkinson's disease patients receiving a Peloton indoor cycle and a heart rate monitor strap delivered to the home, and asked to cycle 3x/week for 12 months with goal of progressing to 45 minute sessions with the heart rate monitor at an aerobic intensity between 60-80% of heart rate reserve with a target cadence between 80-90 revolutions per minute (RPMs). Participants also receive and are asked to wear activity monitors throughout the day to monitor daily. activity levels. Participants also receive biweekly telephone calls to review electronic activity monitoring and exercise data, monitor falls and adverse events, and for guidance on progressing their cycling exercise sessions. See Alberts JL et al., Physical Therapy, 2021;101:1-10.
- Usual and Customary Care Group: Mild to moderate Parkinson's disease patients receiving no active exercise intervention through the research. These participants continued to receive usual and customary care (UCC) for their Parkinson's disease during the 12 month follow-up period. Participants receive and are asked to wear activity monitors throughout the day to monitor daily activity levels, and not to commence a cycling exercise program for the duration of the 12 month follow-up period. Participants also receive biweekly telephone calls to review electronic activity monitoring data, monitor falls and adverse events, and to provide them similar contact time as for the active exercise group.
- Total: Total of all reporting groups
Arm/Group | High-Intensity Aerobic Exercise Group | Usual and Customary Care Group | Total
Number analyzed (Participants) | 129 | 127 | 256
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 70 | 53 | 123
  >=65 years | 59 | 74 | 133
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.1 (8.6) | 65.2 (8.2) | 64.2 (8.5)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Sex/Prefer not to answer | 1 | 0 | 1
  Male | 86 | 84 | 170
  Female | 42 | 43 | 85
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 2 | 6
  Not Hispanic or Latino | 125 | 125 | 250
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 1 | 4
  White | 123 | 121 | 244
  More than one race | 1 | 3 | 4
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 129 | 127 | 256
Movement Disorder Society-Unified Parkinson's Disease Rating Scale (Motor Examination) [Mean (Standard Deviation); unit: units on a scale] — Movement Disorder Society Unified Parkinson's Disease Rating Scale Part III: Motor Examination score, measured off medication. Range of scores is 0 to 132, with lower score indicating better motor function. Population: All observed data are summarized; 5 participants, 3 in the aerobic exercise (AE) and 2 in the usual care (UC) arm, withdrew prior to initiating randomized treatment and follow-up, of whom 4 had not yet completed the baseline MDS-UPDRS III. One participant was withdrawn by the study PI due to periodic atrial fibrillation, 2 withdrew due to COVID-19 pandemic-related logistical issues and safety concerns, and 2 withdrew due to dissatisfaction with their randomized usual care assignments.
  units on a scale
    number analyzed (Participants) | 127 | 125 | 252
    (all) | 38.5 (15.6) | 36.9 (14.2) | 37.7 (14.9)
Clinical Site [Count of Participants; unit: Participants]
  Cleveland Clinic | 66 | 65 | 131
  University of Utah | 63 | 62 | 125

OUTCOME MEASURES:

1. Primary Outcome: Movement Disorder Society Unified Parkinson's Disease Rating Scale Part III: Motor Examination Score
Description: Movement Disorder Society Unified Parkinson's Disease Rating Scale Part III: Motor Examination score, measured off medication. Range of scores is 0 to 132, with lower score indicating better motor function.
Time Frame: Baseline, 6 months, 12 months
Population: Means and standard deviations are for the observed data, without imputation of missing data due to baseline or subsequent dropouts. Analytic modeling results reported below are based on the full intention-to-treat population, with missing data multiply-imputed.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Aerobic Exercise Group | Usual and Customary Care Group
Number analyzed (Participants) | 129 | 127
Score on a scale
  Baseline: number analyzed (Participants) | 127 | 125
  Baseline | 38.5 (15.6) | 36.9 (14.2)
  6 months: number analyzed (Participants) | 125 | 123
  6 months | 35.9 (14.1) | 38.8 (15.7)
  12 months: number analyzed (Participants) | 123 | 123
  12 months | 37.1 (13.7) | 40.5 (16.4)
Statistical Analysis 1: Comparison: Aerobic Exercise Group vs Usual and Customary Care Group; Linear mixed model for baseline, 6 month, and 12 month data, with fixed effects of clinical site, treatment, and linear time nested in treatment arm, and AR(1) covariance structure, fit by residual pseudolikelihood maximization (RSPL) in SAS PROC GLIMMIX; Test type: Superiority; p < 0.0001, Mixed Models Analysis — This was the sole primary outcome. The test was conducted with a priori p-value threshold of α=0.05, with no multiple comparison adjustment; Test of equality of slopes with time (change in points/year) between aerobic exercise (AE) and usual and customary care (UCC) treatment arms; Difference in slopes. = -3.62, 95% CI 2-sided [-5.40 to -1.85], Standard Error of Mean 0.91 — Higher MDS-UPDRS III score reflects worse Parkinson's symptoms; increases reflect PD progression. The reported effect is the estimated difference between annual rates of change in scores of AE and UCC patients

2. Secondary Outcome: 10 Meter Walk Test (10MWT) Comfortable Pace Velocity
Description: The 10 Meter Walk Test (10MWT) evaluates gait speed similarly in separate trials with the participant instructed to walk at comfortable and fast pace, and velocity timed over the middle six meters. This outcome is the velocity (meters/second) with instructions to walk at a comfortable pace, performed off medication. Higher velocities indicate better motor function.
Time Frame: Baseline, 6 months, 12 months
Population: Medians and interquartile ranges are for the observed data, without imputation of missing data due to baseline or subsequent dropouts. Analytic results reported below are based on the full intention-to-treat population, with missing data multiply-imputed.
Measure: Median (Inter-Quartile Range); unit: meters/second
Arm/Group | Aerobic Exercise Group | Usual and Customary Care Group
Number analyzed (Participants) | 129 | 127
meters/second
  Baseline: number analyzed (Participants) | 127 | 125
  Baseline | 1.22 [1.07 to 1.39] | 1.26 [1.10 to 1.38]
  6 months: number analyzed (Participants) | 125 | 122
  6 months | 1.23 [1.09 to 1.39] | 1.25 [1.08 to 1.36]
  12 months: number analyzed (Participants) | 121 | 118
  12 months | 1.24 [1.08 to 1.39] | 1.24 [1.06 to 1.38]
Statistical Analysis 1: Comparison: Aerobic Exercise Group vs Usual and Customary Care Group; Linear mixed model for baseline, 6 month, and 12 month data, with fixed effects of clinical site, treatment, and linear time nested in treatment arm, and compound symmetry covariance structure, fit by residual pseudolikelihood maximization (RSPL) in SAS PROC GLIMMIX. To reduce skew and better meet modeling assumptions, test velocity was squared ((meters/second)^2) for modeling. Study sample size was based on the primary outcome, and power was not calculated for this and other outcomes; Test type: Superiority — Equality of annual slopes in squared 10 Meter Walk Test Comfortable Pace Velocity for the AE and UCC groups; p = 0.043, Mixed Models Analysis — Family-wise error controlled at α=0.05 by Holm-Bonferroni adjustment for other motor domain secondary outcomes: 10 Meter Walk Test fast pace velocity, TUG duration & turning velocity, Manual Dexterity Test; Difference in squared velocity slopes = 12.07, 95% CI 2-sided [3.10 to 21.32], Standard Error of Mean 4.65 — The reported effect is the difference in annual slope of meters^2/second, in 100ths of meters^2/second/year. The confidence interval is not multiple comparison adjusted. Parkinson's progression limits mobility; higher slope reflects less progression

3. Secondary Outcome: 10 Meter Walk Test (10MWT) Fast Pace Velocity
Description: The 10 Meter Walk Test (10MWT) evaluates gait speed similarly in separate trials with the participant instructed to walk at comfortable and fast pace, and velocity timed over the middle six meters. This outcome is the velocity (meters/second) with instructions to walk at a fast pace, performed off medication. Higher velocities indicate better motor function.
Time Frame: Baseline, 6 months, 12 months
Population: Means and standard deviations are for the observed data, without imputation of missing data due to baseline or subsequent dropouts. Analytic results reported below are based on the full intention-to-treat population, with missing data multiply-imputed.
Measure: Mean (Standard Deviation); unit: meters/second
Arm/Group | Aerobic Exercise Group | Usual and Customary Care Group
Number analyzed (Participants) | 129 | 127
meters/second
  Baseline: number analyzed (Participants) | 127 | 125
  Baseline | 1.66 (0.34) | 1.67 (0.33)
  6 months: number analyzed (Participants) | 125 | 122
  6 months | 1.67 (0.35) | 1.64 (0.36)
  12 months: number analyzed (Participants) | 121 | 118
  12 months | 1.67 (0.36) | 1.64 (0.39)
Statistical Analysis 1: Comparison: Aerobic Exercise Group vs Usual and Customary Care Group; Linear mixed model for baseline, 6 month, and 12 month data, with fixed effects of clinical site, treatment, and linear time nested in treatment arm, and heterogeneous compound symmetry covariance structure, fit by residual pseudolikelihood maximization (RSPL) in SAS PROC GLIMMIX; Test type: Superiority — Equality of annual slopes in 10 Meter Walk Test Fast Pace Velocity for the AE and UCC groups; p = 0.48, Mixed Models Analysis — Family-wise error controlled at α=0.05 by Holm-Bonferroni adjustment for other motor domain secondary outcomes: 10 meter walk test comfortable pace, Timed Up and Go Test duration and turning velocity, Manual Dexterity Test; Difference in slopes = 3.16, 95% CI 2-sided [-2.10 to 8.42], Standard Error of Mean 2.68 — The reported effect is the difference in annual slopes of the AE and UCC treatment arms, in 100ths of meters/second/year. The confidence interval is not multiple comparison adjusted. Higher slope reflects less Parkinson's disease progression

4. Secondary Outcome: Timed Up and Go (TUG) Test Duration
Description: iPad-facilitated Timed Up and Go Test duration, measured off medication. The Timed "Up & Go" (TUG) Test requires an individual to (1) stand from a chair, (2) ambulate 3 m, (3) turn 180 degrees, (4) ambulate back to the chair, and (5) turn and sit. To perform an instrumented TUG, an Apple iPad is attached to the individual's waist (sacral level) via an adjustable belt. This outcome is the total time to complete this test, in seconds, measured off medication. Lower times indicate better motor function.
Time Frame: Baseline, 6 months, 12 months
Population: Medians and interquartile ranges are reported for the observed data, without imputation of missing data due to baseline or subsequent dropouts. Analytic modeling results reported below are based on the full intention-to-treat population, with missing data multiply-imputed.
Measure: Median (Inter-Quartile Range); unit: seconds
Arm/Group | Aerobic Exercise Group | Usual and Customary Care Group
Number analyzed (Participants) | 129 | 127
seconds
  Baseline: number analyzed (Participants) | 127 | 125
  Baseline | 9.9 [8.5 to 11.7] | 10.0 [8.6 to 11.7]
  6 months: number analyzed (Participants) | 125 | 122
  6 months | 10.4 [8.7 to 11.5] | 10.3 [8.9 to 12.0]
  12 months: number analyzed (Participants) | 121 | 116
  12 months | 9.9 [8.7 to 11.9] | 10.3 [8.8 to 12.1]
Statistical Analysis 1: Comparison: Aerobic Exercise Group vs Usual and Customary Care Group; Linear mixed model for baseline, 6 month, and 12 month data, with fixed effects of clinical site, treatment, and linear time nested in treatment arm, and compound symmetry covariance structure, fit by residual pseudolikelihood maximization (RSPL) in SAS PROC GLIMMIX. To reduce skew and better meet modeling assumptions, test duration was inverted to TUG completions/second. Sample size was based on the primary outcome, and power was not calculated for this and other outcomes; Test type: Superiority — Equality of annual slopes of inverse Timed Up and Go Test duration, i.e., of TUG completions/second, the speed of completing the test; p = 0.16, Mixed Models Analysis — Family-wise error controlled at α=0.05 by Holm-Bonferroni adjustment for other motor domain secondary outcomes: 10 meter walk test comfortable & fast pace, Timed Up and Go Test turning velocity, and Manual Dexterity Test; Difference between estimated annual slopes in TUG completions/second/year for the AE and UCC groups; Difference in slopes = 4.04, 95% CI 2-sided [0.20 to 7.89], Standard Error of Mean 1.96 — Timed Up and Go test speed is expected to decline with Parkinson's progression. The reported effect is the difference between estimated annual slopes for the AE and UCC groups in 1000ths of a TUG completion/second/year

5. Secondary Outcome: Timed Up and Go (TUG) Test Turning Velocity
Description: iPad-facilitated Timed Up and Go Test mean turning velocity, measured off medication. The Timed "Up & Go" (TUG) Test requires an individual to (1) stand from a chair, (2) ambulate 3 m, (3) turn 180 degrees, (4) ambulate back to the chair, and (5) turn and sit. To perform an instrumented TUG, an Apple iPad is attached to the individual's waist (sacral level) via an adjustable belt. This outcome is the mean velocity during performance of step (3), turn 180 degrees, in degrees/second, measured off medication. Higher turn velocities indicate better motor function.
Time Frame: Baseline, 6 months, 12 months
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: degrees/second
Arm/Group | Aerobic Exercise Group | Usual and Customary Care Group
Number analyzed (Participants) | 127 | 125
degrees/second
  Baseline | 77.3 (19.0) | 78.5 (16.6)
  6 months: number analyzed (Participants) | 125 | 122
  6 months | 76.3 (18.0) | 74.5 (18.6)
  12 months: number analyzed (Participants) | 121 | 116
  12 months | 77.1 (18.5) | 76.8 (18.9)
Statistical Analysis 1: Comparison: Aerobic Exercise Group vs Usual and Customary Care Group; Linear mixed model for baseline, 6 month, and 12 month data, with fixed effects of clinical site, treatment, and linear time nested in treatment arm, and compound symmetry covariance structure, fit by residual pseudolikelihood maximization (RSPL) in SAS PROC GLIMMIX. Study sample size was based on the primary outcome, and power was not calculated for this and other outcomes; Test type: Superiority — Test of equality of average turning velocities; p = 0.69, Mixed Models Analysis — Family-wise error controlled at α=0.05 by Holm-Bonferroni adjustment for other motor domain secondary outcomes: 10 meter walk test comfortable & fast pace, Timed Up and Go Test duration, and Manual Dexterity Test; Difference in slopes. = 1.85, 95% CI 2-sided [-1.17 to 4.88], Standard Error of Mean 1.54 — Timed Up and Go test speed is expected to decline with Parkinson's progression. The reported effect is the difference between estimated annual slopes of average turning velocity for the AE and UCC groups in degrees/second/year

6. Secondary Outcome: Manual Dexterity Test Completion Time
Description: Manual Dexterity Test time to completion in seconds, measured off medication. This test is an electronic (iPad-based), modified version of the 9-hole peg test, where an individual is required to grasp, transfer, and release pegs into a 3×3 grid. Participants are asked to grasp and place pegs into holes, and then to return them to their starting locations, as rapidly as possible. Completion times for two repetitions conducted with each hand were averaged. Shorter completion times indicate better motor function.
Time Frame: Baseline, 6 months, 12 months
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: Time (seconds) to completion
Arm/Group | Aerobic Exercise Group | Usual and Customary Care Group
Number analyzed (Participants) | 129 | 127
Time (seconds) to completion
  Baseline: number analyzed (Participants) | 127 | 125
  Baseline | 26.4 [22.7 to 30.2] | 26.1 [23.7 to 29.1]
  6 months: number analyzed (Participants) | 125 | 121
  6 months | 26.4 [23.9 to 30.3] | 26.0 [23.7 to 29.4]
  12 months: number analyzed (Participants) | 120 | 118
  12 months | 26.1 [23.2 to 30.3] | 26.5 [23.0 to 29.7]
Statistical Analysis 1: Comparison: Aerobic Exercise Group vs Usual and Customary Care Group; Linear mixed model for baseline, 6 and 12 month data, with fixed effects of clinical site, treatment, and linear time nested in treatment arm, and compound symmetry covariance structure, fit by residual pseudolikelihood maximization (RSPL) in SAS PROC GLIMMIX. To reduce skew and better meet modeling assumptions, test duration was transformed for modeling to peg transfers/second (18/seconds). Sample size was based on the primary outcome, and power was not calculated for this and other outcomes; Test type: Superiority — Test of equality of slopes of test performance speed (peg transfers/second/year) for AE and UCC groups; p = 0.72, Mixed Models Analysis — Family-wise error controlled at α=0.05 by Holm-Bonferroni adjustment for other motor domain secondary outcomes: Timed Up and Go Test (TUG) duration & turning velocity and 10 meter walk test comfortable & fast pace; Difference in slopes. = -3.62, 95% CI 2-sided [-23.68 to 16.45], Standard Error of Mean 10.23 — Manual dexterity expressed as peg transfers/second is expected to decline with Parkinson's progression. The reported effect is the difference between estimated annual slopes for the AE and UCC groups in 1000ths of a peg transfer/second/year

7. Secondary Outcome: Processing Speed Test Match Score
Description: The Processing Speed Test is a self-administered electronic (iPad) facilitated symbol-number matching task that is similar to the Symbol Digital Modalities Test. Participants are shown a table with numerical labels for 9 disparate symbols, and a second table with a row of such symbols and a blank row beneath it, and asked to complete the second table with the numbers from the first table corresponding to each symbol in the second. When the table is completed, additional tables are shown. The response recorded is the number of correct matches of symbols with numbers in 120 seconds, measured off medication. Higher values indicate faster neural processing.
Time Frame: Baseline, 6 months, 12 months
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: Correct symbol/number matches
Arm/Group | Aerobic Exercise Group | Usual and Customary Care Group
Number analyzed (Participants) | 129 | 127
Correct symbol/number matches
  Baseline: number analyzed (Participants) | 124 | 125
  Baseline | 45.0 [39.0 to 51.0] | 44.0 [38.0 to 49.0]
  6 month: number analyzed (Participants) | 124 | 123
  6 month | 46.0 [37.5 to 51.0] | 45.0 [37.0 to 49.0]
  12 month: number analyzed (Participants) | 122 | 117
  12 month | 44.0 [37.0 to 53.0] | 45.0 [37.0 to 53.0]
Statistical Analysis 1: Comparison: Aerobic Exercise Group vs Usual and Customary Care Group; Linear mixed model for baseline, 6 month, and 12 month data, with fixed effects of clinical site, treatment, and linear time nested in treatment arm, and heterogeneous compound symmetry covariance structure, fit by residual pseudolikelihood maximization (RSPL) in SAS PROC GLIMMIX. To reduce skew and better meet modeling assumptions, test duration was squared (matches^2) for analysis. Study sample size was based on the primary outcome, and power was not calculated for this and other outcomes; Test type: Superiority — Test of equality of slopes of squared match scores (matches^2/year) between AE and UCC groups; p = 0.48, Mixed Models Analysis — Family-wise error controlled at α=0.05 by Holm-Bonferroni adjustment for other non-motor domain secondary outcomes: Visual Memory Test and Trail Making Test B to A duration ratio; Difference in slopes. = -96.91, 95% CI 2-sided [-232.41 to 38.60], Standard Error of Mean 69.12 — Processing speed is expected to decline with Parkinson's, hence duration of the test to increase. The reported effect is the difference in annual slopes (matches^2/year) between the AE and UCC treatment arms

8. Secondary Outcome: Trail Making Test (TMT) B to A Duration Ratio
Description: Participants completed iPad versions of Trail Making Tests A and B (TMT A and B, respectively), with durations in seconds recorded for each. TMT A, considered predominantly a motor task, requires the participant to use a stylus to connect dots in ascending numeric order (1-2-3-4 . . . ). The TMT B, requires the participant to connect dots in an ascending and alternating alpha and numeric order (1-A-2-B . . . .). The total times to complete each of the TMT A and B tasks are automatically recorded by the iPad. This outcome is the (unitless) ratio of the duration to complete Trail Making Test B to the duration to complete Trail Making Test A, reflecting the cognitive burden of visual attention and set-switching, measured off medication. Higher values reflect greater relative burden of the additional cognitive component.
Time Frame: Baseline, 6 months, 12 months
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: unitless ratio
Arm/Group | Aerobic Exercise Group | Usual and Customary Care Group
Number analyzed (Participants) | 129 | 127
unitless ratio
  Baseline: number analyzed (Participants) | 125 | 125
  Baseline | 1.58 [1.22 to 1.93] | 1.55 [1.23 to 2.11]
  6 months: number analyzed (Participants) | 121 | 122
  6 months | 1.51 [1.19 to 2.14] | 1.52 [1.19 to 2.11]
  12 months: number analyzed (Participants) | 118 | 116
  12 months | 1.44 [1.14 to 1.79] | 1.52 [1.21 to 1.98]
Statistical Analysis 1: Comparison: Aerobic Exercise Group vs Usual and Customary Care Group; Linear mixed model for baseline, 6 month, and 12 month data, with fixed effects of clinical site, treatment, and linear time nested in treatment arm, and compound symmetry covariance structure, fit by residual pseudolikelihood maximization (RSPL) in SAS PROC GLIMMIX. To reduce skew and better meet modeling assumptions, the ratios were transformed to their natural logarithms for modeling. Study sample size was based on the primary outcome, and power was not calculated for this and other outcomes; Test type: Superiority — Test of equality of annual slopes of log(TMT B to TMT A duration ratio) for AE and UCC groups; p = 1.00, Mixed Models Analysis — Family-wise error controlled at α=0.05 by Holm-Bonferroni adjustment for other non-motor domain secondary outcomes: Processing Speed Test and Visual Memory Test; Difference in slopes = -3.42, 95% CI 2-sided [-15.31 to 8.46], Standard Error of Mean 6.06 — Visual attention and set switching speed decline with Parkinson's, hence duration of Trail Making Test B increases. The reported effect is the difference in annual slopes of (log TMT B/TMT A), i.e., change/year, between AE and UCC treatment arms

9. Secondary Outcome: Visual Memory Test Symbol Recall Score
Description: Electronics-based test of episodic memory performed on an iPad, reported as number of correctly recalled symbols arrayed on a grid, with values ranging from 0 to 70 and higher numbers reflective of better memory, measured off medication.
Time Frame: Baseline, 6 months, 12 months
Population: Medians and quartiles are for the observed data, without imputation of missing data due to baseline or subsequent dropouts. Analytic modeling results reported below are based on the full intention-to-treat population, with missing data multiply-imputed.
Measure: Median (Inter-Quartile Range); unit: Number correct
Arm/Group | Aerobic Exercise Group | Usual and Customary Care Group
Number analyzed (Participants) | 129 | 127
Number correct
  Baseline: number analyzed (Participants) | 127 | 125
  Baseline | 49 [39 to 59] | 48 [35 to 58]
  6 month: number analyzed (Participants) | 125 | 123
  6 month | 56 [43 to 64] | 54 [44 to 62]
  12 month: number analyzed (Participants) | 122 | 119
  12 month | 57.5 [46 to 63] | 52 [45 to 62]
Statistical Analysis 1: Comparison: Aerobic Exercise Group vs Usual and Customary Care Group; Linear mixed model for baseline, 6 month, and 12 month data, with fixed effects of clinical site, treatment, and linear time nested in treatment arm, and compound symmetry covariance structure, fit by residual pseudolikelihood maximization (RSPL) in SAS PROC GLIMMIX. To reduce skew and better meet modeling assumptions, the score was squared for statistical modeling. Sample size was based on the primary outcome, and power was not calculated for this and other outcomes; Test type: Superiority — Test of equality of annual slopes of squared test score; p = 0.91, Mixed Models Analysis — Family-wise error controlled at α=0.05 by Holm-Bonferroni adjustment for other non-motor domain secondary outcomes: Processing Speed Test and Trail Making Test Ratio; Difference in slopes = 0.16, 95% CI 2-sided [-2.58 to 2.91], Standard Error of Mean 1.40 — Visual memory declines with Parkinson's, hence the score declines. The reported effect is the difference in annual slopes, i.e., changes in mean score^2/year, for AE and UCC treatment arms, shown in hundreds. Higher slope indicates slower decline

ADVERSE EVENTS:
Time Frame: 12 Months
Arm/Group | Aerobic Exercise Group | Usual and Customary Care Group
All-Cause Mortality (participants affected / at risk) | 0/129 | 0/127
Serious Adverse Events (participants affected / at risk) | 10/129 | 15/127
Other Adverse Events (participants affected / at risk) | 27/129 | 0/127
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Aerobic Exercise Group (N=129) | Usual and Customary Care Group (N=127)
Cardiac Disorders (Cardiac disorders) | 1 | 2
Gastrointestinal disorders (Gastrointestinal disorders) | 1 | 1
Infections and infestations (Infections and infestations) | 2 | 3
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 2 | 4
Psychiatric disorder (Psychiatric disorders) | 1 | 0
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Surgical and medical procedure (Surgical and medical procedures) | 3 | 2
Musculoskeletal and connective tissue disorder (Musculoskeletal and connective tissue disorders) | 1 | 1
Nervous System Disorder (Nervous system disorders) | 1 | 2
Renal and urinary disorders (Renal and urinary disorders) | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Aerobic Exercise Group (N=129) | Usual and Customary Care Group (N=127)
Musculoskeletal and Connective Tissue Disorders (Musculoskeletal and connective tissue disorders) | 27 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2021-11-09): https://cdn.clinicaltrials.gov/large-docs/60/NCT04000360/Prot_000.pdf
  • Statistical Analysis Plan (2024-01-29): https://cdn.clinicaltrials.gov/large-docs/60/NCT04000360/SAP_001.pdf
  • Informed Consent Form (2021-12-28): https://cdn.clinicaltrials.gov/large-docs/60/NCT04000360/ICF_002.pdf